CLINICAL TRIAL: NCT02681692
Title: Effect of Magnetic Endoscopic Imaging on Patient Pain During Colonoscopy: a Randomized, Controlled Trial Using a Simple Colon Force Measurement Device
Brief Title: Effect of Magnetic Endoscopic Imaging on Patient Pain During Colonoscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Zhizheng Ge, Director of digestive endoscopy center of Renji hospital, Shanghai Jiao Tong University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: rj（2015）086k
Record Dates: First submitted 2016-02-10; First posted 2016-02-12 (Estimated); Last update posted 2018-07-02 (Actual); Status verified 2018-06

CONDITIONS: Colonic Diseases
Keywords: colonoscopy; colonoscopy education; magnetic endoscope imaging; Colonic Diseases
MeSH Terms: conditions — Colonic Diseases

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- MEI colonoscopy Group (Active Comparator): Patients would be randomly assigned to have colonoscopy examination performed by one inexperienced colonoscopist (having performed less than 200 procedures) with the assistance of magnetic scope navigation system
  Interventions: Device: Magnetic endoscopic imaging system
- Standard colonoscopy Group (No Intervention): Patients would be randomly assigned to have colonoscopy examination performed by one inexperienced colonoscopist (having performed less than 200 procedures) without the assistance of magnetic scope navigation system
- MEI colon model Group (Active Comparator): Colonoscopist would be randomized to perform colonoscopy on a colon model with an MEI view while the force measurement device being used to collect data of colon force variation meanwhile. No patients would be involved in this part.
  All force variation data would be recorded by a image storage device.
  Interventions: Device: Magnetic endoscopic imaging system
- Standard colon model Group (No Intervention): Colonoscopist would be randomized to perform conventional colonoscopy on a colon model without an MEI view while the force measurement device being used to collect data of colon force variation meanwhile. No patients would be involved in this part. All force variation data would be recorded by a image storage device.

INTERVENTIONS:
Device: Magnetic endoscopic imaging system — In the first part,patients would be randomly assigned to have colonoscopy examination performed by one inexperienced colonoscopist (having performed less than 200 procedures) with the assistance of magnetic scope navigation system In the second part colonoscopist would be randomized to perform conventional colonoscopy on a colon model with an MEI view while the force measurement device being used to collect data of colon force variation meanwhile. No patients would be involved in this part. All force variation data would be recorded by a image storage device.
  Other Names: magnetic scope navigation system.; MEI system
  Arms: MEI colon model Group; MEI colonoscopy Group

SUMMARY:
Colonoscopy is widely considered as the main choice for patients with suspected colorectal disease,and for screening those at high risk of colorectal cancer. However， colonoscope examination,especially those unsedated ones for screening,may bring much pain to patients,even induce some severe complications such as perforation.Considering the increasing need of colonoscopy examination for screening purpose,it has been a problem deserving of further study that how to reduce pain and ensure safety during the procedure.Some studies suggest that use of Magnetic endoscopic imaging(MEI) during colonoscopy has the potential to ease patient discomfort and reduce complications.Theoretically,the MEI could accurately depict the position of the scope in three dimensions and help avoid forcefully feeding the colonoscope through loops of vulnerable bowel,thus alleviating patient pain and promoting procedure safety.However,the problem whether MEI system could help reduce patient pain during procedure effectively，especially in inexperienced colonoscopists，still remains controversial for researchers,and no study has been designed to test the hypothesis that MEI may help decrease the risk of some complications,such as colon perforation.In this study we aim to evaluate the he efficacy of magnetic scope navigation on patient pain during unsedated colonoscopy；In addition，we try to construct a simple colon force measurement device ,and by using this device to observe the variation of force exerted on colon loop ,we expect to find the potential mechanism of pain-alleviation and explore the possible effect of complication reduction during colonoscopy under the influence of MEI system.

DETAILED DESCRIPTION:
This clinical trial is planned as two parts:In the first part,consecutive patients would be recruited and randomized to have colonoscopy examination performed by inexperienced colonoscopists (having performed less than 200 procedures) either with or without the assistance of magnetic scope navigation system. The second part would be conducted as a pilot study,we would first construct a simple colon force measurement device;then colonoscopist would be randomized to perform colonoscopy on a colon model either with or without an MEI view while the force measurement device being used to collect data of colon force variation meanwhile. All force variation data would be recorded by a image storage device.No patients would be involved in the second part.In this pilot study, we plan to perform 40 colonoscopy procedures with the assistance of MEI and 40 colonoscopy procedures without the assistance of MEI.

ELIGIBILITY:
Inclusion Criteria:

colonoscopists: All colonoscopists are selected from the colonoscopy learners in Endoscopy Center of Shanghai Renji Hospital. Only inexperienced colonoscopists (having performed less than 200 procedures) would be allowed to participate in the first part while both inexperienced colonoscopists and experienced colonoscopists (having performed less than 350 procedures) are allowed to participate in the second part.

patients: in the first part: Patients aged between 18 and 75 are recruited to receive unsedated colonoscopy examination with their permission. Written informed consent would be obtained.

in the second part:no patient would participate in this part

Exclusion Criteria： patients:consecutive patients,excluding inpatients,pregnant,who had a known or suspected colonic stricture or obstruction, who had previous history of abdominal surgery,who had severe comorbid cardiopulmonary,kidney,liver conditions,who had pacemakers or internal defibrillators,who were unable to give informed consent,who have active gastrointestinal bleeding are recruited

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 594 (Actual)
Dates: Start 2016-04; Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
patients over pain experience | day of colonoscope performance
  A pain score would be obtained from patients shortly after each examination. The score would be obtained with the Help of a visual analogue scale ranging from 0(no pain)to10(the worst pain).
Maximum target colon loop force | day of colonoscope performance
  In the second part,The maximum colon force exerted on a chosen target colon loop （we plan to choose one loop of sigmoid colon）would be recorded by the simple colon force measurement device.

SECONDARY OUTCOMES:
number of attempts of abdominal hand pressure | day of colonoscope performance
number of patient reposition | day of colonoscope performance
endoscopist perception of ease of procedure | day of colonoscope performance
  Endoscopist are asked to score the ease of each procedure after completion,using a ten-point scoring system(ease-of-procedure score)form 0(easiest)to 10(most difficult).
patient's intention to attend unsedated colonoscopy again | day of colonoscope performance
  patients need to answer "yes"or"no"
caecal intubation rate | one year
  Criteria for reaching the caecum are identification of the ileocaecal valve
caecal intubation time | day of colonoscope performance
ime for the colonoscopist to advance to splenic flexure of colon | day of colonoscope performance
  In the second part，time for the colonoscopist to advance to splenic flexure of colon would be recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Gastroenterology, Renji Hospital, Shanghai Institute of Digestive Diseases, Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Background] Continuing Medical Education Exam: September 2014 James Buxbaum, MD, William Ross, MD, Shou-Jiang Tang, MD, Brian Weston, MD,Co-Editors, CME Section G. S. Raju, MD,Editor, CME Section Glenn M. Eisen, MD, MPH,Editor-in-Chief, Gastrointestinal Endoscopy 503.e1， GASTROINTESTINAL ENDOSCOPY Volume 80, No. 3 : 2014
- [Background] Hoff G, Bretthauer M, Dahler S, Huppertz-Hauss G, Sauar J, Paulsen J, Seip B, Moritz V. Improvement in caecal intubation rate and pain reduction by using 3-dimensional magnetic imaging for unsedated colonoscopy: a randomized trial of patients referred for colonoscopy. Scand J Gastroenterol. 2007 Jul;42(7):885-9. doi: 10.1080/00365520601127125. PMID 17558914
- [Background] Shah SG, Brooker JC, Williams CB, Thapar C, Saunders BP. Effect of magnetic endoscope imaging on colonoscopy performance: a randomised controlled trial. Lancet. 2000 Nov 18;356(9243):1718-22. doi: 10.1016/S0140-6736(00)03205-0. PMID 11095259
- [Background] Kaltenbach T, Leung C, Wu K, Yan K, Friedland S, Soetikno R. Use of the colonoscope training model with the colonoscope 3D imaging probe improved trainee colonoscopy performance: a pilot study. Dig Dis Sci. 2011 May;56(5):1496-502. doi: 10.1007/s10620-011-1614-1. Epub 2011 Mar 16. PMID 21409379